CLINICAL TRIAL: NCT00312091
Title: A Phase I/II Comparative Pharmacokinetic Study of the Fixed-Dose Combination (FDC) of Stavudine (d4T), Lamivudine (3TC), and Nevirapine (NVP) as GPO-VIR Pediatric Chewable Tablets Versus the Individual Liquid Formulations in HIV Infected Children 6 Months and Older to Less Than 13 Years of Age in Thailand
Brief Title: Drug Levels of Tablet and Liquid Forms of Lamivudine, Nevirapine, and Stavudine in HIV Infected Thai Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P1056; 10139 (Registry Identifier: DAIDS ES); PACTG P1056; IMPAACT P1056
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Pharmacokinetics; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Lamivudine; Nevirapine; Stavudine; Tablets; stavudine, lamivudine, nevirapine drug combination

ARMS (4):
- A, Stage 1 (Experimental): Tablet containing d4T, 3TC, and NVP taken orally twice daily for the first 4 weeks, then liquid formulations of d4T, 3TC, and NVP taken orally twice daily for the final 4 weeks
  Interventions: Drug: Lamivudine, nevirapine, and stavudine fixed-dose tablet; Drug: Lamivudine; Drug: Nevirapine; Drug: Stavudine
- A, Stage 2 (Experimental): Tablet containing d4T, 3TC, and NVP taken orally twice daily for 4 weeks, then liquid formulations of d4T, 3TC, and NVP taken orally twice daily for 4 weeks
  Interventions: Drug: Lamivudine, nevirapine, and stavudine fixed-dose tablet; Drug: Lamivudine; Drug: Nevirapine; Drug: Stavudine
- B, Stage 1 (Experimental): Liquid formulations of d4T, 3TC, and NVP taken orally twice daily for 2 weeks, then tablet containing d4T, 3TC, and NVP taken orally twice daily for 2 weeks
  Interventions: Drug: Lamivudine, nevirapine, and stavudine fixed-dose tablet; Drug: Lamivudine; Drug: Nevirapine; Drug: Stavudine
- B, Stage 2 (Experimental): Liquid formulations of d4T, 3TC, and NVP taken orally twice daily for 4 weeks, then tablet containing d4T, 3TC, and NVP taken orally twice daily for 4 weeks
  Interventions: Drug: Lamivudine, nevirapine, and stavudine fixed-dose tablet; Drug: Lamivudine; Drug: Nevirapine; Drug: Stavudine

INTERVENTIONS:
Drug: Lamivudine, nevirapine, and stavudine fixed-dose tablet — 7 mg d4T, 30 mg 3TC, 50 mg NVP tablet
  Other Names: GPO-Vir; d4T/3TC/NVP
Drug: Lamivudine — Dosage dependent on weight. More information on this criterion can be found in the protocol.
Drug: Nevirapine — Dosage dependent on weight. More information on this criterion can be found in the protocol.
Drug: Stavudine — Dosage dependent on weight. More information on this criterion can be found in the protocol.

SUMMARY:
The purpose of this study is to compare the blood levels, absorption, and breakdown of lamivudine (3TC), nevirapine (NVP), and stavudine (d4T) in a fixed-dose tablet to that of the individual liquid formulations of the same anti-HIV drugs in HIV infected Thai children.

DETAILED DESCRIPTION:
The Thai Ministry of Public Health strives to provide the HIV infected people of Thailand with affordable antiretrovirals (ARVs). A fixed-dose combination tablet of 3TC, NVP, and d4T is recommended as first-line treatment in HIV infected adults in Thailand. There has been no similar product developed for children for several reasons: pediatric dosing is based on age, weight, or body surface area; developmental changes may influence the bioavailability and pharmacokinetics (PK) of ARVs; and medication adherence may also be a problem. The purpose of this study is to gather bioavailability and PK data in children taking a fixed-dose tablet of 3TC, NVP, and d4T. This information will then be compared to the bioavailability and PK of the individual liquid formulations of these ARVs.

This study has two stages. Stage 1 will last a minimum of 4 weeks; Stage 2 will last a minimum of 8 weeks. In Stage 1, patients will be randomly assigned to one of two arms. Arm A will receive the fixed-dose tablet twice daily for 2 weeks, then switch to the individual liquid formulations twice daily for 2 weeks. Arm B will receive the individual liquid formulations twice daily for 2 weeks, then switch to the fixed-dose tablet twice daily for 2 weeks. To encourage medication adherence, study staff will make home visits and phone calls to each patient's parent or guardian the first week of each treatment regimen. Medical history, a physical exam, and urine collection will occur on Days 11 and 25. Also on Days 11 and 25, patients will be admitted to the hospital to ensure 100% medication adherence and to provide blood for PK studies.

Stage 1 patients are not eligible for Stage 2. In Stage 2, patients will be stratified by body weight, then randomly assigned to one of two arms. Arm A will receive the fixed-dose tablet twice daily for 4 weeks, then switch to the individual liquid formulations twice daily for 4 weeks. Arm B will receive the individual liquid formulations twice daily for 4 weeks, then switch to the fixed-dose tablet twice daily for 4 weeks. To encourage medication adherence, study staff will make home visits and phone calls to each patient's parent or guardian the first week of each treatment regimen. Medical history, documentation of direct observation of therapy (DOT), a physical exam, and urine collection will occur on Days 25 and 53. Also on Days 25 and 53, patients will be admitted to the hospital to ensure 100% medication adherence and to provide blood for PK studies.

ELIGIBILITY:
Inclusion Criteria for Stages 1 and 2:

* HIV infected
* On a highly active antiretroviral regimen (HAART) including NVP and 2 nucleoside reverse transcriptase inhibitors and receiving a maintenance of NVP for at least 4 weeks prior to study entry and taking the current recommended oral dose every 12 hours
* Willing to swallow or chew study drugs
* Willing to be hospitalized for the 12 hour PK studies
* Willing to use acceptable forms of contraception
* Parent or guardian willing to provide informed consent

Inclusion Criteria for Stage 1:

* Between 12 to 30 kg (26.5 to 66.1 lbs)

Inclusion Criteria for Stage 2:

* Between 6 to 30 kg (13.2 to 66.1 lbs)

Exclusion Criteria:

* Certain abnormal laboratory values
* Require certain medications
* Grade 2 or greater vomiting within 30 days prior to study entry
* Grade 2 or greater diarrhea within 30 days prior to study entry
* History of immunological failure (CD4 percentage decrease of more than 30% within a 6-month period for children 6 years or younger OR CD4 cell count decrease of more than 30% within a 6-month period for children older than 6 years)
* Current treatment for acute serious bacterial, viral, or opportunistic infection
* History of dose-limiting toxicity requiring treatment discontinuation of any of the study drugs
* Known hypersensitivity to any of the study drugs
* Current surgical or medical problem affecting gastrointestinal motility or absorption (e.g., ileus, ulcerative colitis) or liver function
* Treatment with immune modulators or myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic, or cytotoxic drugs within 30 days prior to study entry. Patients who have received therapeutic vaccines are not excluded.
* Treatment with experimental drugs within 30 days of study entry
* Acute inflammation of the liver
* Chemotherapy for active cancer
* Any clinically significant diseases other than HIV infection or clinically significant findings that, in the investigator's opinion, may interfere with the study
* Inability to provide a reliable means of contact (e.g., telephone number)
* Pregnancy

Ages: 6 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2006-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Comparative bioavailability | Throughout study
therapeutic adequacy | Throughout study

SECONDARY OUTCOMES:
Drug absorption from standard pharmacokinetic (PK) analyses | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Nirun Vanprapar, MD, Study Chair — Pediatric Infectious Unit, Department of Pediatrics, Siriraj Hopstial, Mahidol University
Locations (4):
- Thailand (4):
  - Queen Sirikit National Institute of Child Health, Pediatric Infectious Unit, Bangkok, Ratchathewi
  - Siriraj Hospital Mahidol University CRS, Bangkok, Ratchathewi
  - Chiang Mai University Pediatrics-Obstetrics CRS, Chiang Mai
  - Chonburi Hosp. CRS, Chonburri

REFERENCES:
- [Background] Chokephaibulkit K, Plipat N, Cressey TR, Frederix K, Phongsamart W, Capparelli E, Kolladarungkri T, Vanprapar N. Pharmacokinetics of nevirapine in HIV-infected children receiving an adult fixed-dose combination of stavudine, lamivudine and nevirapine. AIDS. 2005 Sep 23;19(14):1495-9. doi: 10.1097/01.aids.0000183625.97170.59. PMID 16135903
- [Background] Hoody DW, Fletcher CV. Pharmacology considerations for antiretroviral therapy in human immunodeficiency virus (HIV)-infected children. Semin Pediatr Infect Dis. 2003 Oct;14(4):286-94. doi: 10.1053/j.spid.2003.09.004. PMID 14724793
- [Background] King JR, Kimberlin DW, Aldrovandi GM, Acosta EP. Antiretroviral pharmacokinetics in the paediatric population: a review. Clin Pharmacokinet. 2002;41(14):1115-33. doi: 10.2165/00003088-200241140-00001. PMID 12405863
- [Result] Vanprapar N, Cressey TR, Chokephaibulkit K, Muresan P, Plipat N, Sirisanthana V, Prasitsuebsai W, Hongsiriwan S, Chotpitayasunondh T, Eksaengsri A, Toye M, Smith ME, McIntosh K, Capparelli E, Yogev R; IMPAACT P1056 Team. A chewable pediatric fixed-dose combination tablet of stavudine, lamivudine, and nevirapine: pharmacokinetics and safety compared with the individual liquid formulations in human immunodeficiency virus-infected children in Thailand. Pediatr Infect Dis J. 2010 Oct;29(10):940-4. doi: 10.1097/INF.0b013e3181e2189d. PMID 20453709